CLINICAL TRIAL: NCT02989948
Title: Safety and Effectiveness of Physician-Modified Fenestrated and Branched Aortic Endografting for the Treatment of Thoracoabdominal Aortic Aneurysms (TAAA)
Brief Title: Physician-Modified Fenestrated and Branched Aortic Endografting for TAAA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, David Kuwayama, Associate Professor of Surgery, Yale University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D18194; 2000035699 (Other: Yale IRB)
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Aortic Aneurysm, Thoracoabdominal
Keywords: endovascular; physician-modified; graft; fenestration
MeSH Terms: conditions — Aortic Aneurysm, Thoracoabdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Main Arm - Physician-modified fenestrated endovascular graft (Experimental): Use of a physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft for the endovascular treatment of asymptomatic, non-ruptured thoracoabdominal aortic aneurysms of any Crawford extent (I-V) meeting traditional size criteria for open surgical repair.
  Interventions: Device: Physician-modified aortic endograft
- Expanded Access Arm - Physician-modified fenestrated endovascular graft. (Experimental): Use of a physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft for the endovascular treatment of asymptomatic, non-ruptured thoracoabdominal, thoracic, or abdominal aortic aneurysms of any Crawford extent (I-V) meeting traditional size criteria for open surgical repair in an expanded use population.
  Interventions: Device: Physician-modified aortic endograft

INTERVENTIONS:
Device: Physician-modified aortic endograft — Use of physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft for the endovascular treatment of asymptomatic, non-ruptured thoracoabdominal aortic aneurysms of any Crawford extent (I-V) meeting traditional size criteria for open surgical repair.

SUMMARY:
The primary clinical objective of this study is to evaluate the safety and effectiveness of a physician-modified, fenestrated and branched aortic endoprosthesis for the treatment of thoracoabdominal aortic aneurysms (TAAAs). The goal of the primary analysis is to demonstrate both the safety and effectiveness of using a physician-modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft as compared to previously published results of open surgical replacement of the aneurysmal aorta.

DETAILED DESCRIPTION:
This study is a prospective, two-arm, traditional feasibility study of a physician modified fenestrated Cook Zenith Alpha Thoracic Endovascular Graft base device in adult patients meeting traditional size criteria for open surgical treatment of thoracoabdominal aortic aneurysms (TAAAs). Patients meriting surgical treatment of their aneurysm that also meet inclusion and exclusion criteria will be eligible for enrollment. Patients will be followed for 5 years post procedure. Major adverse events (MAEs) will also be recorded by the Sponsor-Investigator (S-I) and will be monitored by a locally appointed Data Monitoring Committee, Dartmouth-Hitchcock Health and the D-HH Human Research Protection Program IRB/IEC, and the FDA. This record was transferred to Yale in October 2024.

ELIGIBILITY:
MAIN ARM - Inclusion Criteria:

1. Must be a man or woman 50 years of age or older by the date of informed consent.
2. Must have a thoracoabdominal aortic aneurysm of any Crawford classification (extent I-V) that extends no more proximal than the left subclavian artery.
3. Must have an aneurysm size that meets standard indications for surgical repair (6.0 cm in maximum diameter in the descending thoracic aorta, or 5.5 cm in maximum diameter in the abdominal aorta).
4. Must be considered, in the judgment of the S-I, to be a high risk candidate for open surgical repair.
5. Must not be a candidate for repair under the Instructions for Use of a commercially available, FDA-approved endovascular graft.
6. Must be able to provide informed consent.
7. Must be able to comply with the five year study assessment schedule of events.
8. Must have a non-aneurysm-related life expectancy, in the judgment of the S-I, of greater than 2 years.

MAIN ARM - Exclusion Criteria:

1. Aneurysm due to acute or chronic dissection, intramural hematoma, penetrating aortic ulceration, pseudoaneurysm, mycotic aneurysm, or traumatic transection.
2. Ruptured or acutely symptomatic aortic aneurysm.
3. Known connective tissue disorder.
4. Imaging demonstrating any of the following:

   * Lack of 20 mm non-aneurysmal proximal seal zone (zone 3, or zone 2 with a carotid-subclavian bypass or transposition).
   * Lack of 15 mm non-aneurysmal distal seal zone(s) (aortic, common iliac, or external iliac).
   * Branch vessel target (renal, superior mesenteric, or celiac) < 5 mm or > 10 mm in average diameter.
   * Untreated left subclavian artery stenosis or occlusion.
   * Untreated unilateral or bilateral hypogastric artery occlusion.
   * Signs that the inferior mesenteric artery is indispensable.
   * Have branching, duplication, aneurysm, or untreatable stenosis of the celiac, superior mesenteric artery, or renal arteries that would preclude implantation of the investigational devices.
5. Known sensitivities or allergies to stainless steel, PTFE, polyester, polypropylene, nitinol, or gold.
6. History of anaphylaxis to contrast, with inability to prophylax appropriately.
7. Have uncorrectable coagulopathy.
8. Have unstable angina.
9. Have a body habitus that would inhibit X-ray visualization of the aorta.
10. Have a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned ≤30 days of the endovascular repair.
11. Known to be participating in any other clinical study which may affect performance of this device.
12. Known, visible, or suspected pregnancy, confirmed with a Urine Pregnancy Test (UPT)
13. Contraindication to oral antiplatelet therapy.
14. Prisoners or those on alternative sentencing.
15. Known systemic infection with potential for endovascular graft infection.
16. Anticipated need for MRI scanning within 3 months of insertion of investigational product.
17. Other conditions or comorbidities that, in the opinion of the S-I, would exclude the patient.

EXPANDED ACCESS ARM - Inclusion Criteria

1. Must be a man or woman 50 years of age or older by the date of informed consent
2. Must have a thoracic, thoracoabdominal, or abdominal aortic aneurysm that necessitates coverage of one or more visceral vessels (celiac, superior mesenteric, or renals) for establishment of proximal and/or distal seal.
3. Must have an aneurysm size that meets standard size indications for surgical repair (6.0 cm in maximum diameter in the descending thoracic aorta, or 5.5 cm in maximum diameter in the abdominal aorta); or, in the judgment of the S-I, has aneurysm characteristics that portend a high risk of near-term rupture
4. Must be considered, in the judgement of the S-I, to be a high risk candidate for open surgical repair
5. Must not be a candidate for repair under the Instructions for Use of a commercially available, FDA-approved endovascular graft
6. Patient must be able to provide informed consent
7. Must be able to comply with the five year study assessment schedule of events
8. Must have a non-aneurysm-related life expectancy, in the judgement of the S-I, of greater than 2 years

EXPANDED ACCESS ARM - Exclusion Criteria

1. Known or suspected mycotic aneurysm
2. Ruptured aneurysm with hemodynamic instability
3. Known connective tissue disorder
4. Imaging demonstrating any of the following:

   * Lack of 20 mm non-aneurysmal proximal seal zone (in either native aorta, elephant trunk graft, or aortic arch endograft)
   * Lack of 15 mm non-aneurysmal distal seal zone(s) (in either native aortoiliac vessels, prosthetic aortoiliac grafts, or aortoiliac endografts)
   * Branch vessel target (renal, superior mesenteric, or celiac) > 10 mm in average diameter
5. Known sensitivities or allergies to stainless steel, PTFE, polyester, polypropylene, nitinol, or gold
6. History of anaphylaxis to contrast, with inability to prophylax appropriately.
7. Have uncorrectable coagulopathy
8. Have a body habitus that would inhibit X-ray visualization of the aorta
9. Have a major surgical or interventional procedure unrelated to the treatment of the aneurysm planned ≤ 30 days of the endovascular repair
10. Known to be participating in any other clinical study which may affect performance of this device
11. Known, visible, or suspected pregnancy, confirmed with a Urine Pregnancy Test (UPT)
12. Contraindication to oral antiplatelet therapy
13. Prisoners or those on alternative sentencing
14. Known systemic infection with potential for endovascular graft infection
15. Anticipated need for MRI scanning within 3 months of insertion of investigational product
16. Other conditions or comorbidities that, in the opinion of the S-I, would exclude the patient

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-04-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
30 day survival | 30 Days
  Percent of patients who survive 30 days following surgery
Major Adverse Events (MAE) at 30 days following surgery | 30 Days
  Percent of patients who development major adverse events
Treatment success at 12 months following surgery | 12 Months
  Percent of patients achieving treatment success through 1 year
Technical success at 12 months following surgery | 12 Months
  Technical success is assessed 12 months following surgery and is defined as a composite of: successful delivery, without need for unanticipated corrective intervention related to delivery; successful and accurate deployment at the intended implantation site; and successful withdrawal, without need for unanticipated correct intervention related to withdrawal.

SECONDARY OUTCOMES:
Technical success on the day of surgery | Day of Surgery
  Percent of patients achieving technical success on the day of surgery, defined as the composite of; successful delivery, successful and accurate deployment, successful withdrawal.
Aneurysm rupture | Day of Surgery
  Percent of patients developing aneurysm rupture
Conversion to open repair | Day of Surgery
  Percent of patients necessitating conversion to open repair. This is assessed intraoperatively. In case of a device deployment failure or intraoperative aneurysm rupture, emergent conversion to open repair via laparotomy, thoracotomy, or thoracoabdominal aortic exposure may become necessary. Patients undergoing such intraoperative conversion will be considered to have met this endpoint.
Access site complication (Femoral or Iliac) | Day of Surgery
  Percent of patients suffering access site complication (femoral or iliac). If femoral or iliac rupture occurs intraoperatively, or if femoral or iliac flow-limiting dissection or occlusion is identified intraoperatively or on the day of surgery, patients will be considered to have met this outcome.
Lower extremity ischemia | Day of Surgery
  Percent of patients developing lower extremity ischemia. This will be assess intraoperatively and on the day of surgery. If patients have lower extremity pulses either absent or diminished compared to baseline, with associated pain, sensory deficits or motor deficits on clinical evaluation, patients will be considered to have met this outcome.
Lower extremity compartment syndrome | Day of Surgery
  Percent of patients developing lower extremity compartment syndrome. In patients with lower extremity pain to passive motion post-operatively, invasive pressure measurement of the four calf compartments will be performed. If compartment pressures are greater than 30 in any compartment, patients will be considered to have met this outcome.
Stroke | Day of Surgery
  Percent of patients developing stroke - Modified Rankin Score (MRS) of 2 or greater). In patients with altered mental status or lateralizing motor or sensory deficits, MRI of the brain will be performed. If diffusion weighted MRI imaging demonstrates an intracranial lesion, a modified Rankin score will be calculated. If MRS is 2 or greater, patients will be considered to have met this outcome.
Paraplegia | Day of Surgery
  Percent of patients developing paraplegia. Patients with complete absence of lower extremity motor function in one or both legs will be considered to have met this outcome.
Paraparesis | Day of Surgery
  Percent of patients developing paraparesis. Patients will undergo lower extremity motor strength assessment post-operatively on a standard 0 to 5 scale. If greater than 0 but less than 5 in either extremity, patients will be considered to have met this outcome.
Death during surgery | Day of Surgery
  Percent of patients who die during surgery
Survival rate | At 30, 183 days; 1, 2, 3, 4 and 5 years
  Percent of patients who survive
Major Adverse Events (MAEs) | At 30, 183 days; 1, 2, 3, 4 and 5 years
  Percent of patients that development MAEs
Treatment success | At 30, 183 days; 2, 3, 4 and 5 years
  Percent of patients achieving treatment success

CONTACTS AND LOCATIONS:
Overall Officials: David P. Kuwayama, M.D., M.P.A., Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data (IPD) exists at this time.

REFERENCES:
- [Background] Crawford ES, Coselli JS. Thoracoabdominal aneurysm surgery. Semin Thorac Cardiovasc Surg. 1991 Oct;3(4):300-22. No abstract available. PMID 1793767
- [Background] Safi HJ, Miller CC 3rd. Spinal cord protection in descending thoracic and thoracoabdominal aortic repair. Ann Thorac Surg. 1999 Jun;67(6):1937-9; discussion 1953-8. doi: 10.1016/s0003-4975(99)00397-5. PMID 10391343
- [Background] Dapunt OE, Galla JD, Sadeghi AM, Lansman SL, Mezrow CK, de Asla RA, Quintana C, Wallenstein S, Ergin AM, Griepp RB. The natural history of thoracic aortic aneurysms. J Thorac Cardiovasc Surg. 1994 May;107(5):1323-32; discussion 1332-3. PMID 8176976
- [Background] Kuzmik GA, Sang AX, Elefteriades JA. Natural history of thoracic aortic aneurysms. J Vasc Surg. 2012 Aug;56(2):565-71. doi: 10.1016/j.jvs.2012.04.053. PMID 22840907
- [Background] Clouse WD, Hallett JW Jr, Schaff HV, Gayari MM, Ilstrup DM, Melton LJ 3rd. Improved prognosis of thoracic aortic aneurysms: a population-based study. JAMA. 1998 Dec 9;280(22):1926-9. doi: 10.1001/jama.280.22.1926. PMID 9851478
- [Background] Cowan JA Jr, Dimick JB, Henke PK, Rectenwald J, Stanley JC, Upchurch GR Jr. Epidemiology of aortic aneurysm repair in the United States from 1993 to 2003. Ann N Y Acad Sci. 2006 Nov;1085:1-10. doi: 10.1196/annals.1383.030. PMID 17182917
- [Background] O'Callaghan A, Mastracci TM, Eagleton MJ. Staged endovascular repair of thoracoabdominal aortic aneurysms limits incidence and severity of spinal cord ischemia. J Vasc Surg. 2015 Feb;61(2):347-354.e1. doi: 10.1016/j.jvs.2014.09.011. Epub 2014 Oct 23. PMID 25449006
- [Background] Lee JT, Lee GK, Chandra V, Dalman RL. Comparison of fenestrated endografts and the snorkel/chimney technique. J Vasc Surg. 2014 Oct;60(4):849-56; discussion 856-7. doi: 10.1016/j.jvs.2014.03.255. Epub 2014 Apr 27. PMID 24785682
- [Background] Greenberg R, Eagleton M, Mastracci T. Branched endografts for thoracoabdominal aneurysms. J Thorac Cardiovasc Surg. 2010 Dec;140(6 Suppl):S171-8. doi: 10.1016/j.jtcvs.2010.07.061. PMID 21092788
- [Background] Greenberg RK, Lu Q, Roselli EE, Svensson LG, Moon MC, Hernandez AV, Dowdall J, Cury M, Francis C, Pfaff K, Clair DG, Ouriel K, Lytle BW. Contemporary analysis of descending thoracic and thoracoabdominal aneurysm repair: a comparison of endovascular and open techniques. Circulation. 2008 Aug 19;118(8):808-17. doi: 10.1161/CIRCULATIONAHA.108.769695. Epub 2008 Aug 4. PMID 18678769
- [Background] Matsumura JS, Melissano G, Cambria RP, Dake MD, Mehta S, Svensson LG, Moore RD; Zenith TX2 Clinical Trial Investigators. Five-year results of thoracic endovascular aortic repair with the Zenith TX2. J Vasc Surg. 2014 Jul;60(1):1-10. doi: 10.1016/j.jvs.2014.01.043. Epub 2014 Mar 14. PMID 24636714
- [Background] Riga CV, McWilliams RG, Cheshire NJ. In situ fenestrations for the aortic arch and visceral segment: advances and challenges. Perspect Vasc Surg Endovasc Ther. 2011 Sep;23(3):161-5. doi: 10.1177/1531003510388421. Epub 2011 Apr 17. PMID 21502107
- [Background] Oderich GS, Greenberg RK. Endovascular iliac branch devices for iliac aneurysms. Perspect Vasc Surg Endovasc Ther. 2011 Sep;23(3):166-72. doi: 10.1177/1531003511408344. Epub 2011 Aug 1. PMID 21810808
- [Background] Chuter T, Greenberg RK. Standardized off-the-shelf components for multibranched endovascular repair of thoracoabdominal aortic aneurysms. Perspect Vasc Surg Endovasc Ther. 2011 Sep;23(3):195-201. doi: 10.1177/1531003511430397. PMID 22205654
- [Background] Oderich GS, Greenberg RK. The evolving options for endovascular repair of complex aortic aneurysms. Foreword. Perspect Vasc Surg Endovasc Ther. 2011 Sep;23(3):145-8. doi: 10.1177/1531003511407343. No abstract available. PMID 22205653
- [Background] O'Brien N, Sobocinski J, d'Elia P, Guillou M, Maioli F, Azzaoui R, Haulon S. Fenestrated endovascular repair of type IV thoracoabdominal aneurysms: device design and implantation technique. Perspect Vasc Surg Endovasc Ther. 2011 Sep;23(3):173-7. doi: 10.1177/1531003511408340. Epub 2011 Aug 1. PMID 21810817
- [Background] Browne TF, Hartley D, Purchas S, Rosenberg M, Van Schie G, Lawrence-Brown M. A fenestrated covered suprarenal aortic stent. Eur J Vasc Endovasc Surg. 1999 Nov;18(5):445-9. doi: 10.1053/ejvs.1999.0924. PMID 10610834
- [Background] Haulon S, D'Elia P, O'Brien N, Sobocinski J, Perrot C, Lerussi G, Koussa M, Azzaoui R. Endovascular repair of thoracoabdominal aortic aneurysms. Eur J Vasc Endovasc Surg. 2010 Feb;39(2):171-8. doi: 10.1016/j.ejvs.2009.11.009. Epub 2009 Nov 27. PMID 19945316
- [Background] Starnes BW. Physician-modified endovascular grafts for the treatment of elective, symptomatic, or ruptured juxtarenal aortic aneurysms. J Vasc Surg. 2012 Sep;56(3):601-7. doi: 10.1016/j.jvs.2012.02.011. Epub 2012 May 2. PMID 22554425